CLINICAL TRIAL: NCT00149578
Title: A Phase II Study of Induction Chemotherapy Followed by Concurrent Chemotherapy With Radiotherapy in Locally Advanced Pancreatic Cancer
Brief Title: A Phase II Study of Combine Modality Therapy in Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1204
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; gemcitabine; oxaliplatin; 5-Fluorouracil; radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine Oxaliplatin 5FU and Leucovorin

SUMMARY:
Induction chemotherapy will be administered every 2 weeks for 6 cycles (about 3 months). Patients who have radiological evidence of progressive disease will be shifted to salvage chemotherapy. Patients who have responsive or stable disease after induction chemotherapy will receive concurrent chemoradiotherapy 3-4 weeks after the last dose of induction chemotherapy. Surgical evaluation will be performed 4-6 weeks after the completion of chemoradiotherapy. Patients who have resectable disease will undergo surgical resection. Postoperative adjuvant chemotherapy with GOFL for 6 cycles will be given for those who have curative resection. Patients who still have unresectable disease or non-curative resection will receive systemic chemotherapy of GOFL till disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Induction chemotherapy will be administered on a biweekly basis. Reported adverse events and potential risks for gemcitabine, oxaliplatin, 5-FU and leucovorin are described in Section 6. Appropriate dose modifications for are described in Section 5. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

4.1.1 Treatment schedule of induction chemotherapy

For each dose of GOFL chemotherapy, intravenous infusion of gemcitabine at a fixed rate of 10 mg/m2/min will be immediately followed by a 2-hour intravenous infusion of oxaliplatin and then a 48-hour intravenous infusion of 5-FU and leucovorin.

4.1.2 Premedication before chemotherapy

Patients will receive 4mg of dexamethasone and anti-histamine and appropriate anti-emetics (serotonin antagonists) before each dose of chemotherapy.

4.2 Supportive Care Guidelines

Prophylactic G-CSF or GM-CSF will not be routinely used in this study. In case of febrile neutropenia, patients should be treated with appropriate antibiotics. Therapeutic G-CSF may be used at the discretion of attending physicians

4.3 Duration of Induction Chemotherapy

In the absence of treatment delays due to adverse events, treatment may continue for 6 cycles or until one of the following criteria applies:

C Disease progression, C Intercurrent illness that prevents further administration of treatment, C Unacceptable adverse events(s), C Patient decides to withdraw from the study, or C General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

4.4 Agents and Radiation Administration during Concurrent Chemoradiotherapy

4.4.1 Treatment schedule during concurrent chemoradiotherapy

4.4.1.1 Patient selection

Patients were evaluated after 6 cycles of induction chemotherapy. Patients who have progressive disease either due to distant metastasis or locoregional progression will be given salvage systemic chemotherapy and will not be enrolled into concurrent chemoradiotherapy. Patients who achieve complete remission, partial remission or stable disease will be enrolled into 2nd phase of the study, concurrent chemoradiotherapy, 3-4 weeks after the last dose of induction chemotherapy.

4.4.2 Study Agents

Gemcitabine 400mg/m2 will be dissolved in 250ml normal saline and infused intravenously at a fixed rate of 10mg/m2/min for 40 mins.

4.4.1.2 Treatment schedule

Gemcitabine 400mg/m2 in 250ml normal saline will be iv infused for 40mins, 2hrs before RT on day 1, 8, 15, 22, 29, 36. Radiation will be given 180cGy per day, 5 days a week for 28 fractions to totally 5040cGy.

4.4.1.3 Premedication for concurrent chemoradiotherapy

Patients were given dexamethasone 2mg orally three times a day (tid) from the morning of their first radiotherapy fraction. The prophylactic dexamethasone will be continued until after they had received their fifth radiation treatment. Therefore, depending on the day of the week the patients started treatment, dexamethasone will be taken for 5 to 7 days. All patients will be issued with rescue medication, prochlorperazine 10mg every 6 hours orally if they develop nausea and vomiting. If patients still have nausea and/or vomiting during treatment of dexamethasone and prochlorperazine or after the fifth day of radiotherapy, ondansetron 8mg orally or iv one to three times per day or granisetron 1mg per os or iv once everyday 30mins before radiotherapy should be given.

4.4.3 Radiation

4.4.3.1 Radiation technique

Radiation should be performed by high-energy linear accelerators. Three-dimensional radiation treatment planning was used in all cases. Patients will be immobilized in a foam cradle in a supine position, and the treatment planning CT was obtained. Tumor mapping should be performed according to treatment planning CT and the diagnostic CT before induction chemotherapy. Treatment planning was performed with the isocenter calculated at 100% and the 95% line encompassing the planning target volume. The spinal cord was limited to 4600cGy. If one kidney was to receive more than 20Gy then more than 90% of the remaining kidney was excluded from the primary beam. Generally, a three-field no-axial beam arrangement (opposed lateral with an anterior-inferior oblique) was used.

4.4.3.2 Radiation volume

The gross tumor volume is the primary tumor identifiable on CT scan before induction chemotherapy. The clinical target volume was defined as the gross tumor volume plus 0.5cm. The planning target volume was the clinical target volume plus 0.5cm for daily patient set-up variation. No prophylactic nodal irradiation will be given.

4.4.3.3 Radiation dosage

A total dose of 5040cGy in 28 fractions, 180cGy per fraction, one fraction per day, 5 days per week, will be given.

4.5 Surgery

4.5.1 Surgical evaluation

Patients completed induction chemotherapy and concurrent chemoradiotherapy will be evaluated for surgical resection. If there is evidence of distant metastasis, surgery will not be arranged. The feasibility of surgical resection will be evaluated by qualified surgeon according to contrast-enhanced abdominal CT or MRI. Laparoscope is optional for pre-surgical evaluation.

4.5.1.1 Resectable l No distant metastases l Clear fat plane around celiac and superior mesenteric arteries (SMA) l Patent superior mesenteric vein (SMV)/portal vein 4.5.1.2 Borderline resectable l Severe unilateral SMV/portal impingement l Tumor abutment on SMA l Gastroduodenal artery (GDA) encasement up to origin at hepatic artery l Colon or mesocolon invasion l Adrenal, colon or mesocolon, or kidney invasion 4.5.1.3 Unresectable l Distant metastases l SMA, celiac encasement l SMV/portal occlusion l Aortic, inferior vena cava (IVC) invasion or encasement l Invasion of SMV below transverse mesocolon l Rib, vertebral invasion

4.5.2 Treatment schedule of surgery

Surgery will be performed within 4-6 weeks after chemoradiotherapy complete.

4.5.3 Surgical technique

Patients whose tumor are considered to be resectable will undergo laparotomy. If complete surgical resection is feasible, optimal surgery will be performed. If complete surgical resection is impossible, biopsy with or without palliative surgery (eg. bypass surgery) may be performed. 4.6 Adjuvant/Maintenance Chemotherapy

4.6.1 Treatment schedule

Patients who have curative surgical resection will receive 6 cycles of adjuvant GOFL chemotherapy within 4 weeks after surgery and then followed up until tumor progression. Patients who are not feasible for curative resection, will receive continued chemotherapy of GOFL 3-4 weeks after chemoradiotherapy complete. The regimen will continue till disease progression. Patients who develop progressive disease during GOFL will shift to salvage chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of pancreas.
2. Patients must have locally advanced pancreatic cancer.
3. Patients must have unresectable pancreatic cancer evaluated by radiologist and/or surgeon according to either abdominal CT or MRI, or intra-operative findings.

   * Locally advanced unresectable disease was defined by CT or MRI images as low-density tumor (primary and/or lymphadenopathy) with

     1. extension to the celiac axis or superior mesenteric artery,
     2. occlusion of the superior mesenteric-portal venous confluence
     3. aortic, inferior vena cava (IVC) invasion or encasement
     4. invasion of SMV below transverse mesocolon
     5. rib, vertebral invasion
4. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 8.2 for the evaluation of measurable disease.
5. Age >20 years. Because no dosing or adverse event data are currently available on the use of study agents in patients <20 years of age, children are excluded from this study.
6. ECOG performance status 0-2; see Appendix A.
7. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count >1,500/mL
   * platelets >100,000/mL
   * total bilirubin <3X institutional upper limit of normal
   * ALT(SGPT) <5 X institutional upper limit of normal
   * creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
8. Patients who present with jaundice, temporary or permanent internal / external drainage before enrollment will be allowed.
9. The effects of study agents on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with distant metastases are not eligible.
2. Patients may not be receiving any other investigational agents.
3. Patients who have had prior chemotherapy or radiotherapy are not eligible.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents used in the study.
5. Patients who have above grade II peripheral neuropathy.
6. Patients who had non-curable second primary malignancy.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Pregnant women are excluded from this study because the study agents has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
9. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with study agent administered during the study. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2004-10; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to evaluate the local response rate after induction chemotherapy and concurrent chemoradiotherapy in locally advanced pancreatic cancer.
chemotherapy and concurrent chemoradiotherapy in locally advanced pancreatic cancer. .

SECONDARY OUTCOMES:
The secondary end points are to evaluate the distant metastasis rate and time to tumor progression, overall survival time and quality of life after induction

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Ch'ang, M.D., Study Chair — Pancreatic Cancer Disease Committee of Taiwan Cooperative Oncology Group; Li-Tzong Chen, Ph.D., Study Chair — Pancreatic Cancer Disease Committee of Taiwan Cooperative Oncology Group
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District